CLINICAL TRIAL: NCT05550181
Title: Associations of Intraoperative Hypocapnia With Patient Demographics, Ventilation Characteristics and Outcomes--Statistical Analysis Plan for an Individual Patient Data Analysis of PROVHILO and PROBESE
Brief Title: Intraoperative Hypocapnia in PROVHILO and PROBESE
Acronym: iHypoPRO
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Hospital Israelita Albert Einstein (Other); University Hospital Carl Gustav Carus (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Head of the Department, Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: AUMC
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation Complication; Surgery; Pulmonary Complication; Intraoperative Complications; Postoperative Complications
Keywords: Postoperative Complications; Intraoperative Complications; Hypocapnia; Mechanical Ventilation
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications; Hypocapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with hypocapnia: We will use the intraoperatively collected etCO2 levels to classify patients as either 'with hypocapnia' or 'without hypercapnia', using the cutoff of 35 mmHg. A patient is considered 'hypocapnic' if the etCO2 was < 35 mm Hg at any point during surgery, from start of the study till end of the study
  Interventions: Behavioral: intraoperative mechanical ventilation with hypocapnia (etCO2 < 35 mm Hg)
- without hypocapnia: We will use the intraoperatively collected etCO2 levels to classify patients as either 'with hypocapnia' or 'without hypercapnia', using the cutoff of 35 mmHg. A patient is considered 'hypocapnic' if the etCO2 was < 35 mm Hg at any point during surgery, from start of the study till end of the study, and classified as 'without hypocapnia' otherwise. In case of a missing value immediately before extubation, we will use the values as reported in the last hour of surgery.

INTERVENTIONS:
Behavioral: intraoperative mechanical ventilation with hypocapnia (etCO2 < 35 mm Hg) — A patient is considered 'hypocapnic' if the etCO2 was < 35 mm Hg at any point during surgery, from start of the study till end of the study and classified as 'without hypocapnia' otherwise. In case of a missing value immediately before extubation, we will use the values as reported in the last hour of surgery.
  Groups: with hypocapnia

SUMMARY:
To gain a better understanding of the epidemiology of intraoperative hypocapnia, in particular the associations of intraoperative hypocapnia with patient demographics, ventilator characteristics, and perioperative complications we will perform an individual patient-level meta-analysis of two recent randomized clinical trials of intraoperative ventilation, the 'PROtective Ventilation using High versus LOw PEEP trial' (PROVHILO), and the 'Protective intraoperative ventilation with higher versus lower levels of positive end-expiratory pressure in obese patients trial' (PROBESE).

DETAILED DESCRIPTION:
Lung-protective intraoperative ventilation (LPV) has the potential to improve the outcome of surgery patients through a reduction in postoperative pulmonary complications. Use of intraoperative ventilation strategies that use a low tidal volume could result in intraoperative hypercapnia. However, hypocapnia remains surprisingly common during intraoperative ventilation, possibly meaning that anesthesiologists continue to use high, if not too high respiratory rates or tidal volumes.

Previous studies suggested associations between intraoperative derangement of end-tidal carbon dioxide (etCO2) and postoperative outcomes. Indeed, two studies in highly selected patient groups showed associations of intraoperative hypocapnia with prolonged length of hospital stay, in patients undergoing pancreaticoduodenectomy, and in patients undergoing hysterectomy.

To gain a better understanding of the epidemiology of intraoperative hypocapnia, in particular the associations of intraoperative hypocapnia with patient demographics, ventilator characteristics, and perioperative complications we will perform an individual patient-level meta-analysis of two recent randomized clinical trials of intraoperative ventilation; PROVHILO and PROBESE.

ELIGIBILITY:
Inclusion Criteria:

* Planned for major (abdominal) surgery.
* At risk for postoperative pulmonary complications.

Exclusion Criteria:

* Planned thoracic surgery or neurosurgery.
* Unscheduled surgery (i.e., urgent, or emergent surgeries) were excluded because these patients may have had metabolic abnormalities at the moment of surgery, i.e., metabolic acidosis, for which the anesthesiologist may have adjusted the intraoperative ventilator settings. This may have led to a 'compensatory' low etCO2.
* Patients with etCO2 recordings are missing from the study databases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mechanical ventilation for general anesthesia for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2793 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications | Until day seven or hospital discharge, whichever comes first
  Composite of predefined and collected postoperative pulmonary complications. Postoperative pulmonary complications included mild, moderate, and severe respiratory failure; acute respiratory distress syndrome; bronchospasm; new pulmonary infiltrate; pulmonary infection; aspiration pneumonitis; pleural effusions; atelectasis; cardiopulmonary edema; and pneumothorax.

SECONDARY OUTCOMES:
Incidence of intraoperative complications | Intraoperatively
  Defined as intraoperative hypotension, arrhythmias; or need for rescue for desaturations; or need for vasoactive drugs.
Incidence of intensive care unit admission | Until hospital discharge, death or 100 days, whichever comes first
  Incidence of intensive care unit admission during hospital stay
Incidence of extrapulmonary pulmonary complications | Until day seven or hospital discharge, whichever comes first
Incidence of 7-day mortality | Mortality during the first seven days of hospitalization
  Until day seven or hospital discharge, whichever comes first
Incidence of in-hospital mortality | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 days
Incidence of major postoperative complications | Until day seven or hospital discharge, whichever comes first
  Collapsed composite of complications developing within the first seven postoperative combining severe postoperative pulmonary complications, sepsis, septic shock and/or acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Sabrine NT Hemmes, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); David MP van Meenen, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Frederique Paulus, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marcus J Schultz, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Germany
- IRCCS San Martino Policlinico Hospital, Genoa, Italy
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The harmonized dataset will be available after the publication of the main results and under request to the steering committee
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After the publication of the main results

REFERENCES:
- [Background] Deng QW, Tan WC, Zhao BC, Wen SH, Shen JT, Xu M. Intraoperative ventilation strategies to prevent postoperative pulmonary complications: a network meta-analysis of randomised controlled trials. Br J Anaesth. 2020 Mar;124(3):324-335. doi: 10.1016/j.bja.2019.10.024. Epub 2020 Jan 30. PMID 32007240
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Biehl M, Binnekade JM, Canet J, Fernandez-Bustamante A, Futier E, Gajic O, Hedenstierna G, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Putensen C, Ranieri M, Scavonetto F, Schilling T, Schmid W, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network Investigators. Protective versus Conventional Ventilation for Surgery: A Systematic Review and Individual Patient Data Meta-analysis. Anesthesiology. 2015 Jul;123(1):66-78. doi: 10.1097/ALN.0000000000000706. PMID 25978326
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Akkermans A, van Waes JAR, Thompson A, Shanks A, Peelen LM, Aziz MF, Biggs DA, Paganelli WC, Wanderer JP, Helsten DL, Kheterpal S, van Klei WA, Saager L. An observational study of end-tidal carbon dioxide trends in general anesthesia. Can J Anaesth. 2019 Feb;66(2):149-160. doi: 10.1007/s12630-018-1249-1. Epub 2018 Nov 14. PMID 30430440
- [Background] Dony P, Dramaix M, Boogaerts JG. Hypocapnia measured by end-tidal carbon dioxide tension during anesthesia is associated with increased 30-day mortality rate. J Clin Anesth. 2017 Feb;36:123-126. doi: 10.1016/j.jclinane.2016.10.028. Epub 2016 Dec 2. PMID 28183549
- [Background] Dong L, Takeda C, Yamazaki H, Kamitani T, Kimachi M, Hamada M, Fukuhara S, Mizota T, Yamamoto Y. Intraoperative end-tidal carbon dioxide and postoperative mortality in major abdominal surgery: a historical cohort study. Can J Anaesth. 2021 Nov;68(11):1601-1610. doi: 10.1007/s12630-021-02086-z. Epub 2021 Aug 6. PMID 34357567
- [Background] Park JH, Lee HM, Kang CM, Kim KS, Jang CH, Hwang HK, Lee JR. Correlation of Intraoperative End-Tidal Carbon Dioxide Concentration on Postoperative Hospital Stay in Patients Undergoing Pylorus-Preserving Pancreaticoduodenectomy. World J Surg. 2021 Jun;45(6):1860-1867. doi: 10.1007/s00268-021-05984-x. Epub 2021 Feb 16. PMID 33591427
- [Background] Wax DB, Lin HM, Hossain S, Porter SB. Intraoperative carbon dioxide management and outcomes. Eur J Anaesthesiol. 2010 Sep;27(9):819-23. doi: 10.1097/EJA.0b013e32833cca07. PMID 20613537
- [Background] Writing Committee for the PROBESE Collaborative Group of the PROtective VEntilation Network (PROVEnet) for the Clinical Trial Network of the European Society of Anaesthesiology; Bluth T, Serpa Neto A, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE Collaborative Group; Bluth T, Bobek I, Canet JC, Cinnella G, de Baerdemaeker L, Gama de Abreu M, Gregoretti C, Hedenstierna G, Hemmes SNT, Hiesmayr M, Hollmann MW, Jaber S, Laffey J, Licker MJ, Markstaller K, Matot I, Mills GH, Mulier JP, Pelosi P, Putensen C, Rossaint R, Schmitt J, Schultz MJ, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H. Effect of Intraoperative High Positive End-Expiratory Pressure (PEEP) With Recruitment Maneuvers vs Low PEEP on Postoperative Pulmonary Complications in Obese Patients: A Randomized Clinical Trial. JAMA. 2019 Jun 18;321(23):2292-2305. doi: 10.1001/jama.2019.7505. PMID 31157366
- [Background] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] van Meenen DMP, Serpa Neto A, Paulus F, Merkies C, Schouten LR, Bos LD, Horn J, Juffermans NP, Cremer OL, van der Poll T, Schultz MJ; MARS Consortium. The predictive validity for mortality of the driving pressure and the mechanical power of ventilation. Intensive Care Med Exp. 2020 Dec 18;8(Suppl 1):60. doi: 10.1186/s40635-020-00346-8. PMID 33336298
- [Derived] Nasa P, van Meenen DMP, Paulus F, Ferrando C, Bluth T, Gama de Abreu M, Ball L, Bossers SM, Schober P, Schultz MJ, Serpa Neto A, Hemmes SNT; REPEAT; PROVHILO; PROBESE; investigators of the PROVE network; ESAIC CTN. Association of intraoperative end-tidal CO2 levels with postoperative outcomes: a patient-level analysis of two randomised clinical trials. Br J Anaesth. 2025 Dec;135(6):1761-1769. doi: 10.1016/j.bja.2025.07.076. Epub 2025 Sep 10. PMID 40930872

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT05550181/Prot_SAP_000.pdf